CLINICAL TRIAL: NCT04094311
Title: A Phase IIIb Study of the Safety and Efficacy of Tisagenlecleucel Out of Specification for Commercial Release in Patients Who Are Consistent With the Label Indication
Brief Title: Study of Out of Specification for Tisagenlecleucel
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CCTL019B2302
Record Dates: First submitted 2019-09-16; First posted 2019-09-18 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: B-cell Acute Lymphoblastic Leukemia; Diffuse Large B-cell Lymphoma
Keywords: out of specification; tisagenlecleucel; acute lymphoblastic leukemia; large B-cell lymphoma; relapsed/refractory; pediatric; young adult patients
MeSH Terms: conditions — Burkitt Lymphoma; Lymphoma, Large B-Cell, Diffuse; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Recurrence | interventions — tisagenlecleucel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Group A: pALL (Experimental): Pediatric/young adult patients with r/r pALL who meet the indication in the Health Authority-approved CTL019 package insert in the respective country/region whose final manufactured product is OOS for commercial release, but it is considered that the benefit-risk profile may remain favorable and the usual expected benefits of infusing such a product outweigh the potential risks for the patient.
  Interventions: Biological: CTL019
- Group B: r/r LBCL (Experimental): Adult patients with r/r LBCL including DLBCL not otherwise specified, high grade B-cell lymphoma, and DLBCL arising from follicular lymphoma, that is consistent with the Health Authority-approved indication in the package insert for CTL019 in the respective country/region whose final manufactured product is OOS for commercial release, but it is considered that the benefit-risk profile may remain favorable and the usual expected benefits of infusing such a product outweigh the potential risks for the patient.
  Interventions: Biological: CTL019
- Group C: r/r NHL (Experimental): Adult patients with r/r NHL in consistent with the Health Authority approved indication in the package insert for CTL019 in Japan whose final manufactured product is OOS for commercial release, but it is considered that the benefit-risk profile may remain favorable and the usual expected benefits of infusing such a product outweigh the potential risks for the patient.
  Interventions: Biological: CTL019

INTERVENTIONS:
Biological: CTL019 — A single intravenous (i.v.) infusion of CAR-positive viable T cells.
  Other Names: Tisagenlecleucel

SUMMARY:
This study will evaluate the safety of tisagenlecleucel that is out of specification( OOS) for release as commercial product. Specifically, this study will evaluate the safety of CTL019 in the patients treated within the approved label by Japan Health Authority in Part 2. Only for Part 1, in addition to safety, key efficacy of CTL019 will also be evaluated.

DETAILED DESCRIPTION:
This is a single-arm, open-label, multicenter, interventional Phase IIIb study in pediatric/young adult patients with relapsed/refractory (r/r) B-cell acute lymphoblastic leukemia (pALL) and adult patients with r/r large B-cell lymphoma (LBCL) including diffuse large B-cell lymphoma (DLBCL) not otherwise specified, high-grade B cell lymphoma, and DLBCL arising from follicular lymphoma for Part 1 and and r/r ALL and r/r non-Hodgkin's lymphomas (NHL) for Part 2

Patients whose final manufactured tisagenlecleucel patient-specific batch does not meet the approved local commercial release specifications are eligible for inclusion. Each case will be individually assessed and approved by the Novartis manufacturing facility and the Novartis global medical team (including Patient Safety). Following a single infusion of CTL019, the patient will be followed for 3 months for Part 1, and 1 day for Part 2.

ELIGIBILITY:
Key inclusion criteria:

* Signed informed consent/assent must be obtained for this study prior to participation in the study.
* Patients for whom the final manufactured tisagenlecleucel product does not meet the commercial release specifications.
* Not excluded from commercial manufacturing under the Health Authority-approved tisagenlecleucel prescribing information for their respective country/region.
* OOS material has not been deemed to pose an undue safety risk to the patient.
* Patient is suffering from a serious or life-threatening disease or condition.
* Repeat leukapheresis is not clinically appropriate per the investigator assessment.

Key exclusion criteria:

For part 1, patients meeting any of the following criteria are not eligible for inclusion in this study:

* Human immunodeficience virus (HIV) positive patients.
* Patients with active replication of Hepatitis B virus (HBV) or Hepatitis C virus (HCV).
* Patients with primary central nervous system (CNS) lymphoma.
* History of hypersensitivity to any drugs or metabolites of similar chemical classes as tisagenlecleucel.
* Uncontrolled active infection or inflammation.
* Any medical condition identified by the investigator that may impact the assessment of the safety or efficacy outcomes in relation to study treatment.
* Pregnant or nursing (lactating) women. For part 2, exclusion criteria are not set; however, administration should be performed in accordance with the latest versions of the package insert of CTL019.

Ages: 0 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2019-11-21 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Percentage of participants with Adverse Events (AEs) | From Screening up to 3 months for Part 1 and 1 day for Part 2
  Percentage of participants with Serious AEs (SAEs) and non-SAEs

SECONDARY OUTCOMES:
Part 1: Overall Remission Rate in Group A (pALL) | Up to 3 months
  Overall Remission Rate is defined as the percentage of participants wiho achieve a complete remission (CR) and CR with incomplete blood count recovery (CRi) within 3 months following infusion of CTL019 as determined by the local investigator assessment for participants in group A (part 1).
Part 1: Overall Response Rate in Group B (LBCL) | Up to 3 months
  ORR is defined as the percentage of patients who achieve a domplete response and partial response within 3 months following infusion of CTL019 as determined by the local investigator assessment for participants in group B (part 1).

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (47):
- Canada (5):
  - Novartis Investigative Site, Hamilton, Ontario
  - Novartis Investigative Site, Ottawa, Ontario
  - Novartis Investigative Site, Toronto, Ontario
  - Novartis Investigative Site, Montreal, Quebec
  - Novartis Investigative Site, Québec, Quebec
- Japan (42):
  - Novartis Investigative Site, Nagoya, Aichi-ken
  - Novartis Investigative Site, Tōon, Ehime
  - Novartis Investigative Site, Gifu, Gifu
  - Novartis Investigative Site, Sapporo, Hokkaido
  - Novartis Investigative Site, Kobe, Hyōgo
  - Novartis Investigative Site, Nishinomiya, Hyōgo
  - Novartis Investigative Site, Tsukuba, Ibaraki
  - Novartis Investigative Site, Kanazawa, Ishikawa-ken
  - Novartis Investigative Site, Kita-gun, Kagawa-ken
  - Novartis Investigative Site, Yokohama, Kanagawa-ku
  - Novartis Investigative Site, Kyoto, Kyoto
  - Novartis Investigative Site, Tsu, Mie-ken
  - Novartis Investigative Site, Sendai, Miyagi
  - Novartis Investigative Site, Matsumoto, Nagano
  - Novartis Investigative Site, Nagasaki, Nagasaki
  - Novartis Investigative Site, Yufu, Oita Prefecture
  - Novartis Investigative Site, Kurashiki, Okayama-ken
  - Novartis Investigative Site, Izumi, Osaka
  - Novartis Investigative Site, Izumisano, Osaka
  - Novartis Investigative Site, Osaka, Osaka
  - Novartis Investigative Site, Sakai, Osaka
  - Novartis Investigative Site, Suita, Osaka
  - Novartis Investigative Site, Izumo, Shimane
  - Novartis Investigative Site, Hamamatsu, Shizuoka
  - Novartis Investigative Site, Bunkyo Ku, Tokyo
  - Novartis Investigative Site, Bunkyo-ku, Tokyo
  - Novartis Investigative Site, Chuo Ku, Tokyo
  - Novartis Investigative Site, Fuchū, Tokyo
  - Novartis Investigative Site, Minato-ku, Tokyo
  - Novartis Investigative Site, Setagaya-ku, Tokyo
  - Novartis Investigative Site, Shinjuku-ku, Tokyo
  - Novartis Investigative Site, Aomori
  - Novartis Investigative Site, Chiba
  - Novartis Investigative Site, Fukuoka
  - Novartis Investigative Site, Hiroshima
  - Novartis Investigative Site, Kumamoto
  - Novartis Investigative Site, Kyoto
  - Novartis Investigative Site, Niigata
  - Novartis Investigative Site, Okayama
  - Novartis Investigative Site, Osaka
  - Novartis Investigative Site, Saitama
  - Novartis Investigative Site, Wakayama

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com